CLINICAL TRIAL: NCT03894514
Title: Modelo de predicción Multivariable de Resultados de Artroplastia Total de Rodilla
Brief Title: Multi-variable Prediction Model of Total Knee Replacement Outcome
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario La Fe (Other); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: LOS_ATR
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2019-03

CONDITIONS: Knee Osteoarthritis; Joint Disease; Total Knee Replacement; Arthroplasty Complications
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Total knee arthroplasty (TKA) is a surgical procedure applied as a common solution to overcome limitations produced by advanced stages of severe gonarthrosis. The procedure has high prevalence, high associated costs, and is considered to be cost-effective. Rehabilitation is essential to optimize outcomes. However, in clinical practice, the length of rehabilitation for each patient may be highly variable, and the programmed times may lack the necessary objectivity. Current limitation of resources and increasing prevalence make essential to generate strategies to optimize surgical results, so that the use of resources of the health system is efficient without detriment to the patient's benefit. For this purpose, objective and pragmatic information must be available, and should be based on scientific evidence in order to assist in making clinical decisions. Indeed, a number of demographic, biomedical and psychosocial factors have been identified as predictors of TKA results (i.e weight, age, expectations...). Some of them have been associated with the need for hospital resources after surgery. However, most researches base their predictions in retrospective studies, which are limited in the type of variables that can be used (clinic history), quality of registries, and limitations of retrospective designs. On the other hand, most of prospective researches base their predictions in a limited number of outcomes. To overcome this limitations, this project has been designed as a prospective observational study with two observations of each patient.

* The primary goal is to implement a multi-variable prediction model of TKA outcome, so that the procedure become optimal in two aspects : patient recovery (social and economic benefit) and use of health system resources (economic benefit). The implementation requires a processing of the information sampled through various algorithms and innovative data processing in this field, based on data mining and machine learning techniques. This will be used in search of the model with the greatest predictive capacity.
* As a secondary objective, information extracted from patients both in the final stages of the condition, and in the medium term after the intervention will allow to study the functional and psychosocial reality of the subjects with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years old
* Severe knee osteoarthritis
* In the surgery waiting list for undergoing total knee replacement surgery

Exclusion Criteria:

* Lobo Mini-mental State examination < 20 (not able to properly understand the tests and study)
* Vestibular affection that prevents to perform the tests

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe knee osteoarthritis, waiting for total knee replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Length of stay | change from preoperative assessment to six months after surgery
  Length of in-hospital rehabilitation

SECONDARY OUTCOMES:
Oxford knee Score (OKS) | change from preoperative assessment to six months after surgery
  Patient Reported Outcome questionnaire to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty. The OKS consists of twelve questions covering function and pain associated with the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes
International Physical Activity Questionnaires (IPAQ-short form) | change from preoperative assessment to six months after surgery
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives. It consists of open-ended questions surrounding individuals' last 7-day recall of physical activity. Total physical activity is estimated in metabolic (MET) MET-min/week and time spent sitting. Then three level or categories are proposed (1=low, 2=moderate and 3=high level of physical activity)
Euro Quality of Life 5D questionnaire (EQ-5D) | change from preoperative assessment to six months after surgery
  This is a measure of health-related quality of life. The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, with 3 possible answers; the score is obtained from the possible binary combination of answers, and interpreted using the visual analogue scale validation technique for the Spanish population.
Geriatric Depression Scale (GDS) short form | change from preoperative assessment to six months after surgery
  Yesavage Scale. The short form of this questionnaire consists of a 15-item self-report assessment used to identify depression in older adults. Questions are answered "yes" or "no", and results consider and individual to be non depressed (normal<5), probably depressed (mild=5<10) and very likely to ve depressed (severe>10)
Visual Analogue Scale (VAS) of Pain | change from preoperative assessment to six months after surgery
  A visual analog scale is used to assess the perceived knee pain. The participant specifies their level of knee pain by indicating a position along a continuous line between 0, no pain, and 10, worse possible pain
Expectations (Pain and Function) | change from preoperative assessment to six months after surgery
  The individual is asked: "How do you expect to feel after the operation?". The level of expectation is answered with a Likert scale ranging from much worse to much better.
Strength | change from preoperative assessment to six months after surgery
  Quadriceps isometric strength as measured with hand-held dynamometer
Range of Motion | change from preoperative assessment to six months after surgery
  Knee range of motion as measured in degrees with a telescopic goniometer
Timed Up & Go | change from preoperative assessment to six months after surgery
  A timed test used as a measure of mobility and dynamic balance in which the individual raises from an arm-chair, walks three meters, turn round a cone, and go back to sit again
Five times sit to stand test | change from preoperative assessment to six months after surgery
  A measure of physical performance. The functional strength of the lower extremities, the transition movements, the balance and the risk of falls are evaluated. The time spent in getting up from a chair for five times is recorded
One leg balance test | change from preoperative assessment to six months after surgery
  A measure of static balance. The time the patient is able to stand on one leg keeping balance is recorded

OTHER OUTCOMES:
Romberg test (open eyes) | change from preoperative assessment to six months after surgery
  A T-Plate pedometer will be used to register posturographic data. One trial of 30-s with open eyes, in which the individual has to stand over the platform and remain as static as possible during the test. Data extracted include the velocity of center of pressures (in mm/s), the center of pressure excursions (surface in mm2) and weight-bearing data measured as percentage of weight on each leg
Comorbidities | baseline assessment
  Clinical history data of comorbidities (the individual is asked whether other diseases are present, i.e. osteoarthritis in other parts of the body, diabetes, and etc)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia. Facultat de Fisioterapia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided